CLINICAL TRIAL: NCT04090541
Title: Investigating the Immediate Effects of Kinesio Tape and Biomechanical Tape on Strength and Performance: A Randomized Placebo-Controlled Cross-Over Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Mirsad ALKAN, Principal Investigator, Bahçeşehir University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 52
Record Dates: First submitted 2019-08-29; First posted 2019-09-16 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Sports Physical Therapy; Sports Performance
Keywords: Kinesiology Tape; Biomechanical Tape; Performance; Muscle Strength; Vertical Jump

STUDY DESIGN:
Intervention Model Description: This study was conceived as a randomized placebo controlled prospective trial. With the aim of blocking effects of morphological specifities of participants, this study was designed on a four stage application on the same participants. This stages were (1) control testing with No Tape(NT) (2) placebo testing with Sham Tape(ST) application (3) Kinesology Tape(KT) application (4) Biomechanical Tape (BT) application. With the aim of blocking bias effects, randomization was designed with the computerized system using four way algorithm which led to NT, ST, KT and BT applications for each participant in mixed order but all applications have equal time in order.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control (No Intervention): Tests were applied with any taping.
- Sham Taping (Sham Comparator): In ST stage; medical purpose, hypoallergenic OctaCare® Rigid Transparent Plaster was applied as a rigid tape. This tape is also used under rigid tapes for protecting the skin. In this study investigators didn't prefer extra rigid tape on the plaster because that was very light and less sensitive material to our knowledge so it suited our aim of placebo control.
  Interventions: Other: Rigid Tape
- Kinesiology Taping (Experimental): In KT stage; the original Kinesio Tex® Tape Classic was applied as a kinesiology tape. In this study, investigators applied the tape with muscle activation technique and paper of tension (it was declared %10) according to Kenzo Kase's Kinesio Taping concept. It was implemented on both bileral Rectus Femoris and Calf muscles with same technique.
  Interventions: Other: Kinesiology Tape
- Biomechanical Taping (Experimental): In BT stage; Dynamic Tape® was applied as a biomechanical tape. In this study, investigators applied the tape with offload technique and paper of tension according to Ryan Kendrick's Biomechanical Taping concept. It was implemented on both bileral Rectus Femoris and Calf muscles with same technique.
  Interventions: Other: Biomechanical Tape

INTERVENTIONS:
Other: Rigid Tape — Non-Elastic Tape
  Arms: Sham Taping
Other: Kinesiology Tape — Tape can be elongate only one direction
  Arms: Kinesiology Taping
Other: Biomechanical Tape — Tape can be elongate only two direction
  Arms: Biomechanical Taping

SUMMARY:
There has been an increasing interest in Kinesiology Tape(KT) and Biomechanical Tape(BT) in clinics and athletic competitions. Recently; the performance increasing effect of taping methods on healthy subjects in sports is being investigated.

DETAILED DESCRIPTION:
Kinesio Taping (KT) is a technique utilizing a two way elastic tape originally created by Kenzo Kase in the 1970s. KT is a complementary method which is used as an adjunct to major therapy approaches in various musculoskeletal and neurological diseases.4 KT is employed in sports injuries and various health problems; but there is limited scientific evidence evaluating KT effectiveness and the results are inconsistent.5 One of the KT potential benefits is that of raising the range of motion through increasing blood circulation or through stimulation of cutaneous mechanoreceptors and this way it affects fascial tissue.6-8 Biomechanical Taping (BT) is a technique utilizing a four way elastic tape originally created by Ryan Kendrick in the 2010s. BT is a complementary method for supplementing load absorption, force contribution and modifying movement. BT affects tissues and movement in a mechanical way and it is almost a completely different method from KT. Kase's hypothesis is that KT affects fascial tissues and mechanoreseptors, but Kendrick's hypothesis is that BT ,which is applied in shortened position and cross joint segments, will gain potential energy in case of an extremity realized movement with antagonist activity. Then the weak agonist muscle gets activated for repositioning the extremity; this potential energy turns to kinetic energy like a released bow. As a result of kinetic energy, it may support the movement with using passive mechanical strength.9 In this study, the investigators aim to illustrate immediate effects of various taping methods on the performances of healthy subjects. In that way the investigators test hypothesis that different taping methods affect healthy subjects to improve performance. The investigators; investigate strength, active range of motion and vertical jump height as a parameters of performance with No Tape(NT), Sham Tape(ST), KT and BT.

ELIGIBILITY:
Inclusion Criteria:

* 18-24 BMI
* Physically active according to International Physical Activity Questionnarie (IPAQ)

Exclusion Criteria:

* Any known systemic diseases or medical condition
* Sensitive or fragile skin,
* Allergic diseases
* Pregnancy or pregnancy suspicion
* Using of sedative, psychosomatic or analgesic drugs

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
Change From Vertical Jump With Each Taping Application | baseline, and immediate effect in a 15 minutes
  A fotoelectrical sensor base "Micro Gate Opto Jump Next®, software version 1.10, BFS Vertical Jump protocol with three jumps" was used for quantitative analysis of Counter Movement Vertical Jump (CMVJ). Minimum, maximum and average values of jumping height for all jumps (10) were recorded as canti-meter (cm).
Change From Muscle Strength With Each Taping Application | baseline, and immediate effect in a 15 minutes
  A hand held electronic dynamometer "MicroFet® 2" was used to evaluate isometric bilateral knee extension and ankle dorsal flexion strength.11 Measurements were repeated three times and maximum value of strength was recorded as Kilogram-Force (Kg-F).

SECONDARY OUTCOMES:
Change From Active Range Of Motion With Each Taping Application | baseline, and immediate effect in a 15 minutes
  A wide angle webcam "logitech® c920 full hd pro web cam" that was integrated with opto jump software was used for assessment of active range of motion in front of jumping on image based assessment tool of opto jump software. Acromion, Trochantor major of femur, lateral epicondyle of femur, Lateral Condyle of Tibia and medial malleolus of tibia were marked for the indicator before the jumps. Videos, recorded at the same time with jump and synchronous with jumping values, were used for resolving knee and hip flexion degrees before jump with maximum height and they were assessed with indicators on computer surface on optojump software. Values recorded as degrees (º).

CONTACTS AND LOCATIONS:
Overall Officials: Habibe Serap İnal, Principal Investigator — Bahçeşehir University; Şebnem Nur Alkan, Principal Investigator — Bahçeşehir University
Locations (1):
- Bahçeşehir University, Istanbul, Beşiktaş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No